CLINICAL TRIAL: NCT06179459
Title: Registry of Patients Undergoing Endoscopic Management of Pancreatic Fluid Collections
Status: Recruiting | Type: Observational
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 22.060.03
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Acute Pancreatitis; Pancreatic Pseudocyst; Pancreatic Necrosis
MeSH Terms: conditions — Pancreatitis; Pancreatic Pseudocyst; Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic management of pancreatic fluid collections — Patients with pancreatic fluid collections will be undergoing EUS-guided drainage and/or endoscopic necrosectomy

SUMMARY:
Acute pancreatitis is one of the most common gastrointestinal disorders requiring hospitalization worldwide. Pancreatic fluid collections can occur as a consequence of acute and chronic pancreatitis and can result in significant morbidity and mortality, including significant abdominal pain, gastric outlet obstruction, biliary obstruction, organ failure, persistent unwellness, infection and sepsis.

Symptomatic pancreatic fluid collections require treatment, and endoscopic drainage is considered standard of care. The aim of this study is to evaluate the treatment outcomes in patients undergoing standard of care, endoscopic treatment of pancreatic fluid collections.

DETAILED DESCRIPTION:
Acute pancreatitis has an annual incidence of 13-45 cases per 100,000 persons and is one of the most common gastrointestinal disorders requiring hospitalization worldwide. It leads to over a quarter of a million hospital admissions annually in the United States, and inpatient costs exceeding 2.5 billion US dollars. Pancreatic fluid collections can occur as a consequence of acute and chronic pancreatitis and can result in significant morbidity and mortality, including significant abdominal pain, gastric outlet obstruction, biliary obstruction, organ failure, persistent unwellness, infection and sepsis.

Symptomatic pancreatic fluid collections require treatment, and endoscopic drainage is considered standard of care. Endoscopic treatment involves the drainage of the fluid collection into the stomach or duodenum by placement of metal or plastic stents. If clinically indicated, endoscopic necrosectomy is also performed, which is the removal of devitalized pancreatic tissue using the endoscope. Currently the treatment success rate of endoscopic treatment of pancreatic fluid collections exceeds 90%.

The aim of this study is to evaluate the treatment outcomes in patients undergoing standard of care, endoscopic treatment of pancreatic fluid collections.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* All patients undergoing endoscopic treatment of pancreatic fluid collections

Exclusion Criteria:

* Age < 18 years
* Patients who did not receive endoscopic treatment of pancreatic fluid collections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic fluid collections
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Treatment outcomes in patients undergoing endoscopic treatment of pancreatic fluid collections. | 3 years
  Treatment outcomes in patients undergoing endoscopic treatment of pancreatic fluid collections.

SECONDARY OUTCOMES:
Treatment success | 6 months
  Rate of treatment success, defined as the resolution of pancreatic fluid collection on CT scan in association with clinical resolution of symptoms at 6-months from index intervention.
Number and type of interventions performed | 6 months
  Number of interventions performed to achieve treatment success
Need for surgical intervention | 6 months
  Need for any surgical intervention in patients undergoing endoscopic therapy for pancreatic fluid collections.
Technical success of endoscopic interventions in pancreatic fluid collections. | 6 months
  Technical success of endoscopic interventions in pancreatic fluid collections.
Inflammatory response and organ failure in patients undergoing endoscopic therapy for pancreatic fluid collections. | 6 months
  Rate of inflammatory response and organ failure in patients undergoing endoscopic therapy for pancreatic fluid collections.
Disease-related adverse events | 6 monthts
  Rate of disease-related adverse events
Procedure-related adverse events | 6 months
  Procedure-related adverse events in patients undergoing endoscopic management of pancreatic fluid collection
Timing of intervention | 6 months
  Intervention at 4 weeks since onset of pancreatitis (traditional approach) versus intervention when the area of necrosis is contained or only partially encapsulated.
Hounsfield units of the pancreatic fluid collection | 6 months
  Impact of hounsfield units in the necrotic collection on endoscopic intervention
Impact of partial versus full encapsulation of pancreatic fluid collections | 6 months
  Impact of partial versus full encapsulation of pancreatic fluid collections on endoscopic intervention
Incidence of disconnected pancreatic duct syndrome and sequelae of disconnected pancreatic duct syndrome | 3 years
  Incidence of disconnected pancreatic duct syndrome and sequelae of disconnected pancreatic duct syndrome
Hospital admission | 6 months
  Rate of hospital readmissions due to disease-related or procedure-related events in patients undergoing endoscopic therapy for pancreatic fluid collections.
Disease recurrence | 3 years
  Rate of disease recurrence in patients undergoing endoscopic management of pancreatic fluid collections
Diabetes | 3 years
  Rate of diabetes
Exocrine pancreatic insufficiency | 3 years
  Rate of exocrine pancreatic insufficiency

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Bang, MD MPH, Principal Investigator — Orlando Health, Digestive Health Institute
Locations (1):
- Orlando Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No